CLINICAL TRIAL: NCT01679366
Title: The Effectiveness of Probiotics for the Therapy of Acute Pharyngotonsillitis in Adult Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0054-11-ZIV
Record Dates: First submitted 2012-08-16; First posted 2012-09-06 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2011-11

CONDITIONS: Throat Pain
MeSH Terms: conditions — Pharyngitis | interventions — Sugars; Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Penicillin G (No Intervention): hospitalization of 30 patients given penicilline intraveniously for 72 hours
- Placebo (Placebo Comparator): 30 hospitalized patients will be given placebo with a regular penicillin treatment
  Interventions: Drug: Placebo
- Probiotic (Experimental): Probiotics will be given to 30 hospitalized patients with regular penicillin treatment
  Interventions: Drug: Probiotics

INTERVENTIONS:
Drug: Placebo — 1 tablet 2 times daily
  Other Names: Sugar pill for mimic probiotics
  Arms: Placebo
Drug: Probiotics — 1 tablet twice daily
  Other Names: BLIS
  Arms: Probiotic

SUMMARY:
The addition of probiotics to the routine therapy of Acute Pharyngotonsillitis in adult patients may shorten the duration, and reduce the severity of the disease.

DETAILED DESCRIPTION:
Hypothesis The addition of probiotics to the routine therapy of AP in adult patients may shorten the duration, and reduce the severity of the disease.

Study design A prospective, randomized, placebo-controlled, double-blinded study comparing treatment with probiotics to placebo in patients with AP.

The study will be conducted in accordance with the ethical standards of the Helsinki Declaration and will be approved by the Human Experimentation Ethics Committee of the Ziv Medical Center. Signed informed consent will be required from all patients before inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Acute pharyngotonsillitis for which hospitalization for intravenous antibiotic treatment and/or fluids is needed

Exclusion Criteria:

* Current therapy with systemic prednisone or equivalent at 20 mg/d for more than 10 days prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
period of disease | 10 days
  Patients will be followed daily while hospitalized. After discharge patients will fill a daily dairy for 10 days and record symptoms, signs, drinking, eating, and return to normal life. All dairies will be collected on day 10 of the study.

SECONDARY OUTCOMES:
analysis | 10 days
  Follow-up throat culture, CBC, CRP, and ESR on day 4 of the study or at discharge if before. For patients with abnormal laboratory tests on admission, repeat tests are performed before discharge according to the routine of the department. For patients with normal tests on admission, these tests will be part of the study. For patients with Streptococcus pyogenes growth on admission and day 4 of the study, another throat culture will be done on day 10 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Livshits, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv Medical Center, Safed, Israel